CLINICAL TRIAL: NCT02107924
Title: Use of Antibiotic Contained Calcium Sulfate Carrier in Acute Periprosthetic Infections(APPI) of Total Knee Replacements
Brief Title: Use of Antibiotic Carrier in Acute Periprosthetic Infections (APPI) of Total Knee Replacements
Status: Withdrawn | Type: Observational
Why Stopped: No Funding
Sponsor: Michael Muldoon, M.D. (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Michael Muldoon, M.D., Co-Sponsor, Sharp HealthCare
Organization: Sharp HealthCare (Other)
Other Study IDs: 1112-0211
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Infection
Keywords: Total; Knee; Replacment; Infection; Stimulan
MeSH Terms: conditions — Infections | interventions — Stimulan; Tobramycin; Vancomycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- APPI of TKR-Stimulan: Surgery Stimulan beads 2.4 G Tobramycin 2.0 G Vancomycin
  Interventions: Procedure: APPI of TKR-Stimulan
- APPI of TKR-historical: Surgery 2.4 G Tobramycin 2.0 G Vancomycin

INTERVENTIONS:
Procedure: APPI of TKR-Stimulan
  Other Names: Stimulan; Tobramycin; Vancomycin
  Groups: APPI of TKR-Stimulan

SUMMARY:
The purpose of the study is to gather information on the use of Stimulan, the surgery, and anitbiotics to whetether the APPI has decreased or shown improvement when compared to study participants who did not receive Stimulan during their revision total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* APPI within 28 days of primary TKR
* Acute hematogenous infection within 4 weeks of symptoms

Exclusion Criteria:

* Exposed prosthesis
* Infection occuring in revised joints
* Poly articular infections
* have allergies to tobramycin or Vancomycin
* previous chronic infections in or around any ipsilateral extremity trauma or implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total knee replacement and have developed either APPI within 28 dyas of surgery, or an acute onset of a hematogenous (blood-source ) infection in knee, more than 30 days after surgery with symptoms present less than 28 days
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Retention of components | 12 months
Eradication of infection | 12 months

SECONDARY OUTCOMES:
C-Reactive protein (CRP) | 12 months
Wound complications | 12 months
Knee Society Score | 12 months
Visual Analog Scale | 12 months
Outcome Assessment Scores | 12 months
Ongoing use of antibiotics | 6 weeks
AP and lateral Radiographs of involved joint | 12 months
Positive synovial fluid cell count | pre-operative
Sedimentation Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Muldoon, MD, Principal Investigator — Sharp HealthCare; David R Lionberger, MD, Principal Investigator — Southwest Orthopedic Group, LLC
Locations (1):
- Southwest Orthopedic Group, LLP, Houston, Texas, United States

REFERENCES:
- [Background] Parvizi J, Zmistowski B, Berbari EF, Bauer TW, Springer BD, Della Valle CJ, Garvin KL, Mont MA, Wongworawat MD, Zalavras CG. New definition for periprosthetic joint infection: from the Workgroup of the Musculoskeletal Infection Society. Clin Orthop Relat Res. 2011 Nov;469(11):2992-4. doi: 10.1007/s11999-011-2102-9. No abstract available. PMID 21938532
- [Background] Mortazavi SM, Vegari D, Ho A, Zmistowski B, Parvizi J. Two-stage exchange arthroplasty for infected total knee arthroplasty: predictors of failure. Clin Orthop Relat Res. 2011 Nov;469(11):3049-54. doi: 10.1007/s11999-011-2030-8. PMID 21866421
- [Background] Koyonos L, Zmistowski B, Della Valle CJ, Parvizi J. Infection control rate of irrigation and debridement for periprosthetic joint infection. Clin Orthop Relat Res. 2011 Nov;469(11):3043-8. doi: 10.1007/s11999-011-1910-2. PMID 21553171
- [Background] Gardner J, Gioe TJ, Tatman P. Can this prosthesis be saved?: implant salvage attempts in infected primary TKA. Clin Orthop Relat Res. 2011 Apr;469(4):970-6. doi: 10.1007/s11999-010-1417-2. PMID 20544317
- [Background] Estes CS, Beauchamp CP, Clarke HD, Spangehl MJ. A two-stage retention debridement protocol for acute periprosthetic joint infections. Clin Orthop Relat Res. 2010 Aug;468(8):2029-38. doi: 10.1007/s11999-010-1293-9. PMID 20224958